CLINICAL TRIAL: NCT00699244
Title: Selective Local Anesthetic Placement Using Ultrasound-guidance and Neurostimulation for the Infraclavicularbrachial Plexus Block
Brief Title: Comparison of Central Versus Peripheral Placement of Local Anesthetic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Clifford Bowens, Assistant Professor, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 61267
Record Dates: First submitted 2008-06-12; First posted 2008-06-17 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Hand Surgery; Elbow Surgery; Forearm Surgery; Wrist Surgery
Keywords: forearm; hand; elbow; wrist; brachial plexus; infraclavicular block

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peripheral placement of local anesthesia (Experimental): to receive ultrasound guided peripheral placement of local anesthetic
  Interventions: Procedure: Peripheral placement of local anesthesia
- Central placement of local anesthesia (Active Comparator): to receive central placement of local anesthetic
  Interventions: Procedure: Central placement of local anesthesia

INTERVENTIONS:
Procedure: Peripheral placement of local anesthesia — Peripheral placement of local anesthesia
  Arms: Peripheral placement of local anesthesia
Procedure: Central placement of local anesthesia — Central placement of local anesthesia
  Arms: Central placement of local anesthesia

SUMMARY:
Does ultrasound increases the success rate and if there is a difference in success rate between placing the local anesthetic centrally versus peripherally.

DETAILED DESCRIPTION:
A comparison of the infraclavicular placement of local anesthetic either centrally (posterior cord) vs peripheral placement (lateral or medial cord) using ultrasound guidance. This will be done to determine if ultrasound increases the success rate and if there is a difference in success rate between placing the local anesthetic centrally versus peripherally.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) Class I-III.
* Patient is undergoing elective hand or forearm surgery.
* Patient is an adult, 18 years old or older.

Exclusion Criteria:

* Morbid obesity (calculated body mass index > 35 kg/m2).
* Patient unable to cooperate.
* Patient with a known brachial plexus injury.
* Medical contraindication to anesthetic technique (allergy, cardiac condition, neurologic condition, localized infection, bleeding disorder).
* Patients who are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2006-12; Primary Completion 2009-01 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
increase success rate of the block to produce surgical anesthesia and analgesia | during and following surgical procedure

CONTACTS AND LOCATIONS:
Overall Officials: Clifford Bowens, M.D., Principal Investigator — clifford.bowens@vanderbilt.edu
Locations (1):
- Vanderbilt University Orthopedic Surgicenter, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Vanderbilt University Medical Center Department of Anesthesiology — http://www.vandydreamteam.com